CLINICAL TRIAL: NCT05121610
Title: Effects of Different Revascularization Strategies on Cardiovascular Outcomes in Patients With Complex Coronary Artery Disease
Brief Title: Effects of Different Revascularization StrateGies in Complex Coronary Artery DiseasE (EDGE)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, Principal Investigator, Beijing Anzhen Hospital
Other Study IDs: EDGE
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Coronary Artery Disease
Keywords: PCI; CABG; HCR; Complex coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CABG group: CABG group
  Interventions: Procedure: The procedures include PCI, CABG and HCR
- HCR group: HCR group
  Interventions: Procedure: The procedures include PCI, CABG and HCR
- PCI group: PCI group
  Interventions: Procedure: The procedures include PCI, CABG and HCR

INTERVENTIONS:
Procedure: The procedures include PCI, CABG and HCR — The procedures include PCI, CABG and HCR

SUMMARY:
Coronary heart disease is one of the most serious diseases that endanger people's health. Complex coronary artery disease is critical and has high mortality. Therefore, it is urgent to explore the best treatment method for complex coronary artery disease. Some previous studies have shown that patients with left main coronary artery disease with a SYNTAX score> 32 points, and diabetic/non-diabetic three-vessel disease patients with coronary heart disease with a SYNTAX score > 22 points, CABG is recommended for revascularization. However, with the continuous innovation of surgical technology and the rapid development of surgical instruments, the treatment of patients with complex coronary artery disease is increasing. Therefore, it is necessary to investigate the effects of different revascularization strategies on long-term prognosis in patients with complex coronary artery disease (SYNTAX score > 22 points).

ELIGIBILITY:
Inclusion Criteria:

1. Male/female aged 18-80 years;
2. Having complex coronary artery disease (SYNTAX score > 22 points) undergoing myocardial revascularization

Exclusion Criteria:

1. Cardiogenic shock or hemodynamic instability;
2. Undergoing other heart surgery at the same time;
3. Previous coronary artery bypass surgery;
4. History of cerebral hemorrhage;
5. Ischemic stroke in the past six months;
6. History of cancer;
7. Life expectancy no more than 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with complex coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 2864 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
MACCE | 1 year
  Major adverse cardiovascular and cerebrovascular events (MACCE) at 1 year, including all-cause death, non-fatal myocardial infarction, ischemia-driven revascularization, and non-fatal stroke

SECONDARY OUTCOMES:
All cause death | 1 year
  All-cause death is defined as death from cardiovascular causes, death from non-cardiovascular causes, and death from unknown causes.
Cardiovascular death | 1 year
  Cardiovascular death
Non-fatal myocardial infarction | 1 year
  Non-fatal myocardial infarction
Ischemia-driven revascularization | 1 year
  Ischemia-driven revascularization
Non-fatal stroke | 1 year
  Stroke is defined as a neurological deficit with symptoms or signs that last at least 24 hours and imaging studies (CT or MRI) confirm the presence of cerebral infarction or cerebral hemorrhage.
The composite endpoints including all-cause death, non-fatal myocardial infarction, and ischemia-driven revascularization | 1 year
  The composite endpoints including all-cause death, non-fatal myocardial infarction, and ischemia-driven revascularization
The composite endpoints including cardiovascular death, non-fatal myocardial infarction, and non-fatal stroke | 1 year
  The composite endpoints including cardiovascular death, non-fatal myocardial infarction, and non-fatal stroke
The composite endpoints including cardiovascular death or nonfatal myocardial infarction | 1 year
  The composite endpoints including cardiovascular death or nonfatal myocardial infarction
All bleeding events defined by the BARC bleeding criteria | 1 year
  All bleeding events defined by the BARC bleeding criteria
Type 2, 3 and 5 bleeding events defined by the BARC bleeding criteria | 1 year
  Type 2, 3 and 5 bleeding events defined by the BARC bleeding criteria

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Shi, Principal Investigator — Beijing Anzhen Hospital

IPD SHARING:
Plan to Share IPD: Undecided